CLINICAL TRIAL: NCT03437707
Title: Efficacy of Intravenous Ibuprofen and Paracetamol on Postoperative Pain and Morphine Consumption in Lumbar Disc Surgery: Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy of Intravenous Ibuprofen and Paracetamol on Postoperative Pain and Morphine Consumption in Lumbar Disc Surgery
Acronym: ibuprofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sedatakbas2
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain Management
Keywords: Postoperative pain; Intravenous ibuprofen; Intravenous paracetamol; Lumbar disc surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Analgesia, Patient-Controlled; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Placebo-Controlled Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): 250 ml saline will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate
- Intravenous paracetamol (Active Comparator): 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate; Drug: Intravenous paracetamol
- Intravenous ibuprofen (Active Comparator): 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate; Drug: Intravenous ibuprofen

INTERVENTIONS:
Drug: Morphine Sulfate — Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: Intravenous patient-controlled analgesia
Drug: Intravenous paracetamol — 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: paracetamol
  Arms: Intravenous paracetamol
Drug: Intravenous ibuprofen — 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: ibuprofen
  Arms: Intravenous ibuprofen

SUMMARY:
Primary aim of this prospective, randomized, double-blind, placebo-controlled clinical trial is to compare the analgesic effects of IV ibuprofen and paracetamol on postoperative pain, and secondary aim is the effects on morphine consumption and side effects of morphine in patients who underwent lumbar disc surgery with a single level laminectomy or discectomy.

DETAILED DESCRIPTION:
All surgical procedures are associated with acute pain and inflammation, with varying degrees of severity for patients, causing significant stress and discomfort. Effective postoperative pain management in lumbar disc surgery may reduce complications and improve postoperative care. For postoperative pain, multimodal analgesic techniques are used to provide synergistic effects through different nociceptive mechanisms.

Various analgesics are used for pain. Opioids, commonly used for postoperative pain, are the most popular drug group. Side effects such as sedation, respiratory depression, nausea-vomiting, pruritus and urinary retention that develop secondary to opioids may also be reduced by the combination of supplemental analgesics.

Adjuvant agents, including nonsteroidal anti-inflammatory drugs (NSAID), may be used in combination with opioids. These drugs not only reduce pain but also control the underlying inflammatory process. In addition, combining NSAIDs and opioids can help to reduce the side effects by minimizing administration of total opioid consumption.

Intravenous (IV) ibuprofen is the first and only IV NSAID approved in the United States for both pain and fever control in adults. It has been reported in multicenter studies that IV ibuprofen is safe and effective in postoperative pain management for abdominal hysterectomy and orthopedic surgeries.

IV paracetamol is an analgesic and antipyretic agent used as a first step drug for pain and fever control in adults and children. It has been clearly shown that IV paracetamol, with analgesic efficacy and good safety profile, reduces analgesic requirements for pain management. It provides better analgesic efficacy and reduces opioid consumption when used in combination with opioids.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists scores 1-3
* 18-85 years

Exclusion Criteria:

* American Society of Anesthesiologists scores IV,
* Under the age of 18,
* Over the age of 85,
* Peptic ulcer disease,
* Hepatic and renal dysfunction,
* Severe cardiovascular and pulmonary disease,
* Allergic history to propofol, fentanyl, rocuronium, paracetamol, ibuprofen and morphine,
* Emergency surgery,
* Refused informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Visual Analog Scale (VAS, 0-10)

SECONDARY OUTCOMES:
Sedation score | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Ramsey sedation score (1-6)
Morphine consumption | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Morphine

CONTACTS AND LOCATIONS:
Overall Officials: Sedat AKBAS, Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat AKBAS, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tunali Y, Akcil EF, Dilmen OK, Tutuncu AC, Koksal GM, Akbas S, Vehid H, Yentur E. Efficacy of intravenous paracetamol and dexketoprofen on postoperative pain and morphine consumption after a lumbar disk surgery. J Neurosurg Anesthesiol. 2013 Apr;25(2):143-7. doi: 10.1097/ANA.0b013e31827464af. PMID 23360885

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03437707/Prot_SAP_000.pdf